CLINICAL TRIAL: NCT04446026
Title: A Randomized, Placebo-controlled Clinical Trial of Teneligliptin as Quadruple Oral Combination Therapy for Type 2 DM After Failure of an Oral Triple Anti-diabetic Regimen
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 4-2020-0488
Record Dates: First submitted 2020-06-22; First posted 2020-06-24 (Actual); Last update posted 2021-06-09 (Actual); Status verified 2021-06

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — 3-(4-(4-(3-methyl-1-phenyl-1H-pyrazol-5-yl)piperazin-1-yl)pyrrolidin-2-ylcarbonyl)thiazolidine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- teneligliptin (Experimental)
  Interventions: Drug: teneligliptin
- placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: teneligliptin — teneligliptin 20mg PO qd for 24weeks
  Arms: teneligliptin
Drug: Placebo — teneligliptin 20mg PO qd for 12weeks after placebo 1T PO qd for 12 weeks
  Arms: placebo

SUMMARY:
This is a randomized, placebo-controlled clinical trial of Teneligliptin as quadruple oral combination therapy for type 2 diabetes after failure of an oral triple anti-diabetic regimen. Patients with uncontrolled type 2 diabetes (7.1% ≤ HbA1c ≤ 9%) prescribed with triple combination of oral antidiabetic drugs more than 12 weeks with sufficient doses (metformin >= 1000mg/d, Glimepiride >=4 mg/day, Gliclazide >= 60 mg/day, SGLT-2 inhibitor with approved dose by Korea FDA) will be included. Using randomization, patients would take either teneligliptin (20mg) or placebo for 12 weeks. After 12 weeks of trial, all patients would receive teneligliptin for another 12 weeks. As outcomes, changes in HbA1c and fasting plasma glucose at 12th and 24th weeks compared with at baseline, and proportions of patients who achieved a glycemic goal (HbA1c <=7%) at 12th and 24th weeks will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

1. Age over 18 years and less than 81 years
2. Patients with type 2 diabetes prescribed with triple combination of oral antidiabetic drugs more than 12 weeks with sufficient doses (metformin >= 1000mg/d, Glimepiride >=4 mg/day, Gliclazide >= 60 mg/day, SGLT-2 inhibitor with approved dose by Korea FDA)
3. Uncontrolled hyperglycemia with 7.1% ≤ HbA1c ≤ 9% at randomization period
4. Recommended to use insulin by physicians
5. Patients able to understand study protocol and cooperative
6. Voluntary consent to participation of study after understanding study protocol

Exclusion Criteria:

1. Type 1 diabetes, gestational diabetes, other than type 2 diabetes
2. Insulin treatment more than 1 week (not necessarily continuous use) prior to screening visit within 1 year
3. Hypersensitivity to TENELIA tablet including main and other component
4. Use of DPP4 inhibitor more than 1 week prior to screening visit within 3 months or discontinuation of DPP4 inhibitor due to severe side effects regardless of treatment period
5. History of acute or chronic metabolic acidosis and ketosis including diabetic ketoacidosis with/without comma prior to screening visit within 12 weeks
6. Genetic trait of galactose intolerance, Lapp lactase deficiency, or glucose-galactose mal-absorption
7. Difficulty in oral ingestion of drug owing to anatomical abnormalities in head and neck area, or owing to abnormalities in central nervous system
8. Steroid use including per oral and non-oral more than 14 consecutive days prior to screening visit within 8 weeks (inhaled steroid use is permitted)
9. Histories of any malignancy prior to screening visit within 5 years
10. History of congestive heart failure (>= 10) NYHA class III)
11. Uncontrolled arrhythmia, unstable angina, myocardial infarction, stroke, transient ischemic attack, cerebrovascular disease prior to screening visit within 24 weeks
12. Initiation of statin to treat dyslipidemia prior to screening visit within 4 weeks or anticipated increasing dose of statin during study period
13. Renal failure, chronic kidney disease stage <=3 (estimated glomerular filtration rate <30 mL/min/1.73 m2, calculated using EKD-EPI) or patients with dialysis
14. Abnormalities in liver function test: AST, ALT, or ALP >= 2.5 fold of ULN or patients with liver cirrhosis (Child-Pugh class B or C)
15. Infection of HIV, HBV, or HCV and patients subjected to anti-viral therapy within 1 year
16. Pregnant or lactating women; or planning to be pregnant
17. Patients with other severe infection or with severe injuries, or patients expecting any surgery with transient insulin use for peri-operational glucose control
18. Alcohol or any psychotropic substances dependancy , or dependency of any unapproved substances
19. Last visit of other clinical trials for treatment purposes prior to screening visit within 30 days
20. Other inappropriate properties judged by researchers

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2020-07-08 (Actual); Primary Completion 2020-12-07 (Actual); Study Completion 2021-05-17 (Actual)

PRIMARY OUTCOMES:
Hb1Ac | 12 weeks
  Difference between baseline and HbA1c at 12 weeks after treatment with test drug

SECONDARY OUTCOMES:
HbA1c | 24 weeks
  Difference between baseline and HbA1c at 24 weeks after treatment with test drug
Percentage of patients who reached target blood glucose (6.5% or 7% as HbA1c) | 12 weeks
  Percentage of patients who reached target blood glucose (6.5% or 7% as HbA1c) at 12 and 24 weeks after treatment with the test drug
Percentage of patients who reached target blood glucose (6.5% or 7% as HbA1c) | 24 weeks
  Percentage of patients who reached target blood glucose (6.5% or 7% as HbA1c) at 12 and 24 weeks after treatment with the test drug
Fasting glucose | 12 weeks
  Fasting blood glucose (FPG) at 12 and 24 weeks after treatment with test drug
Fasting glucose | 24 weeks
  Fasting blood glucose (FPG) at 12 and 24 weeks after treatment with test drug

CONTACTS AND LOCATIONS:
Locations (1):
- Yonsei Severance Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No